CLINICAL TRIAL: NCT04193267
Title: rTMS for the Improvement of Language Functioning in the Logopenic Variant of Primary Progressive Aphasia; a Feasibility and Tolerability Pilot Study
Brief Title: Can Magnetic Brain Stimulation Improve Language Function in Primary Progressive Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS23339 (B2019:108)
Record Dates: First submitted 2019-11-18; First posted 2019-12-10 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Logopenic Progressive Aphasia
Keywords: Primary Progressive Aphasia; Brain Stimulation
MeSH Terms: conditions — Aphasia, Primary Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): 30 sessions of high-frequency (10Hz) repetitive stimulation applied over the posterior region of the left superior temporal gyrus in patients with logopenic primary progressive aphasia (PPA-L) using a MagStim Rapid2 Transcranial Magnetic Simulation machine.
  Interventions: Device: MagStim Rapid2 Transcranial Magnetic Simulation

INTERVENTIONS:
Device: MagStim Rapid2 Transcranial Magnetic Simulation — A non-invasive method of brain stimulation

SUMMARY:
The purpose of this study is to investigate the feasibility of using repetitive transcranial magnetic stimulation (rTMS) - a form of non-invasive brain stimulation - to improve language functioning in individuals who have the logopenic variant of primary progressive aphasia (PPA-L) - a slowly progressive impairment of language, characterized by difficulties with word-finding, sentence repetition and sentence comprehension.

DETAILED DESCRIPTION:
This study is an open label pilot study that aims to recruit 10 individuals with diagnosed logopenic primary progressive aphasia (PPA-L) to investigate the tolerability and efficacy of using repetitive transcranial magnetic stimulation (rTMS) to improve language functioning in this disorder. rTMS is a non-invasive method of brain stimulation that uses rapid magnetic pulses applied over the scalp to activate neurons in a specified target location of the brain.

A variety of language tests will be administered to participants prior to rTMS treatment as well as following 30 sessions of daily rTMS. Additionally, language testing will be performed during the first session of rTMS treatment in order to assess the effect of simultaneous rTMS administration on language function. Performance on the pre- and post-treatment tests will be compared to determine the effect of rTMS treatment on language abilities.

Treatment will consist of daily sessions of high frequency (10 Hz) rTMS applied over the left temporal gyrus. Patients will receive one session of rTMS per day for 30 consecutive weekdays. Each session will take approximately 45 minutes to complete.

As a pilot study, this research will be used to evaluate the effect size and the feasibility of a more definitive project in the future. Both patient response and tolerability to rTMS will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPA-L (confirmed by a neurologist or neuropsychiatrist who has observed the patient for at least one year);
* Mild to moderate language impairment as assessed by the Druks and Masterson Naming Task;
* Native English speaker.

Exclusion Criteria:

* Cerebrovascular disorders, hydrocephalus or intra-cranial mass, documented by MRI;
* History of traumatic brain injury, seizures, or another neurological disease;
* Significant medical problems (e.g. poorly controlled diabetes or hypertension or cancer within the past 5 years);
* Major depressive disorder, bipolar disorder, schizophrenia, substance use disorder or mental retardation according to the criteria of the DSM-IV;
* Any contraindication for rTMS (e.g., implanted metal devices; cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps, metal in the body [rods, plates, screws, shrapnel, dentures, IUD] or metallic particles in the body, surgical clips in the head, previous neurosurgery, cochlear implants, prosthetic heart valves);
* Currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in score on the Druks and Masterson Naming Task | One week pre- and one week post-rTMS treatment
  Assessment of change in language function as a result of rTMS intervention. Minimum score = 0. Maximum score = 24. Higher scores indicate better naming performance.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Tsang, MD, Principal Investigator — University of Manitoba; Mandana Modirrousta, MD PhD, Study Director — University of Manitoba
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No